CLINICAL TRIAL: NCT01931800
Title: Identification and Quantification of Immune Response Induced by Hyaluronidase and Other Factors of Virulence of Invasive Human Infections of Streptococcus Pneumoniae
Acronym: Hyalo strepto
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: PIROTH PHRC R 2004
Record Dates: First submitted 2013-08-27; First posted 2013-08-29 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Invasive Pneumococcic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Presenting patients a pneumonia pneumococcique
  Interventions: Biological: Sampling of blood
- Patients presenting a bacteremia pneumococcique
  Interventions: Biological: Sampling of blood
- Patients affected by pneumococcique meningitis
  Interventions: Biological: Sampling of blood

INTERVENTIONS:
Biological: Sampling of blood

SUMMARY:
* 4 tubes (2 x7-ml dry tubes with yellow gelose, and 2 x 5 ml tubes with blue CTAD) will be taken from the patient within 24 hours following inclusion (D0) in the department in which the patient is hospitalised
* 4 tubes (2 x7-ml dry tubes with yellow gelose, and 2 x 5 ml tubes with blue CTAD) will be taken from the patient every 7 days following inclusion for 5 weeks (if the patient is still in hospital at the time), in the department where he/she is hospitalised (D7, D14, D21, D28, D35). Samples will no longer be taken once the patient has left the CHU, even if all of the samples have not been taken.
* For children less than 6 years old, only 2 tubes (1 x 7 ml dry tube with yellow gelose, and 1x5 ml tube with blue CTAD) will be taken following the same timetable.
* For hospitalised patients, a leeway of 48 hours is authorized for the sampling procedure. Samples will be taken at the same time samples are taken for the usual care of the patient.
* The tubes will be taken to the Bacteriology Laboratory using the usual collection circuit of the CHU. These tubes will then be redirected to the Infectious Diseases Laboratory to be centrifuged and then stored at -80°C. The strain of Streptococcus pneumoniae isolated in the patient will be preserved at -80°C. If strains other than Streptococcus pneumoniae are isolated, these different strains will all be preserved at -80°C under the same identification number.

ELIGIBILITY:
Inclusion Criteria:

* Patients (children or adults) hospitalised at Dijon CHU
* Presenting invasive pneumococcal disease, confirmed by:

The presence of Streptococcus pneumoniae in a blood culture, or The presence of Streptococcus pneumoniae in a sample of cerebrospinal fluid, or The presence of significant levels of Streptococcus pneumoniae in an endobronchial sample (bronchial brushing or bronchoalveolar lavage), or in protected tracheal aspirations or in the spit of non-hospitalised patients or those in Intensive care Units.

Exclusion Criteria:

- Patients in whom the implication of Streptococcus pneumoniae is suspected because of: positive urinary soluble antigen of Streptococcus pneumoniae with the exclusion of any other positive sample, presence of non- significant levels of Streptococcus pneumoniae in bronchopulmonary samples The presence of significant levels of Streptococcus pneumoniae in protected tracheal aspirations or in the spit, with the exclusion of any other positive sample in patients who had been in an Intensive care Unit for more than 48 hours at the time the sample was taken.

- Patients in whom Streptococcus pneumoniae had already been isolated in the 5 weeks preceding inclusion in the present study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients hospitalized in a service, for whom a sampling "targets" (hémoculture, cerebrospinal fluid, bronchial brush, liquid of broncho-alveolar wash, protected tracheal aspiration) with positive culture to Streptococcus pneumoniae.
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2005-01-06 (Actual); Primary Completion 2015-01-27 (Actual); Study Completion 2015-01-27 (Actual)

PRIMARY OUTCOMES:
Quantification of immune response induced by the hyaluronidase of Streptococcus pneumoniae | In the visit of inclusion then every 7 days during all the duration of patient hospitalization

SECONDARY OUTCOMES:
Quantification of hyaluronidase expression in strains of Streptococcus pneumoniae | In the visit of inclusion then every 7 days during all the duration of his hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon, Dijon, France